CLINICAL TRIAL: NCT06030453
Title: Using SMART HOME Strategy to Reduce the Incidence of Delirium in the Intensive Care Unit: A Randomized Controlled Study
Brief Title: Using SMART HOME Strategy to Reduce the Incidence of Delirium in the Intensive Care Unit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 202307034RIND
Record Dates: First submitted 2023-08-22; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-08

CONDITIONS: Delirium; Intensive Care Unit Delirium
Keywords: The incidence of delirium; The intensive care unit.
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMART HOME Care Gruop (Experimental): Experimental Group:"SMART HOME" refers to a set of interventions aimed at preventing delirium. Sleep hygiene.Multidisciplinary collaboration.Assessment of pain/anxiety/agitation.Release of tracheal tubes and restraints.Time and schedule.Home-like environment and Hearing.Orientation support.Medication review and adjustment.Early mobilization and nutrition.
  Interventions: Combination Product: SMART HOME strategy
- Control Group (Active Comparator): Control Group: The control group will receive traditional comprehensive care in the ICU based on the PADIS (pain, agitation, delirium, immobility, sleep disruption) assessment. This care will be administered by ICU nurses and will include pharmacological treatments for pain, agitation, delirium, immobility, and sleep disruption as well as nursing interventions.
  Interventions: Combination Product: PADIS nursing intervention

INTERVENTIONS:
Combination Product: SMART HOME strategy — Sleep hygiene: quiet and dim environment for 6 hours to facilitate sleep (Score: 0-100%).Multidisciplinary collaboration: pharmacists, respiratory therapists, rehabilitation therapists, and physical therapists (Score: ≥20%).Assessment : Evaluating and assessing the levels of pain, anxiety, and agitation (Score: 0-100%).Release of tracheal tubes and restraints: relieving pressure from tracheal tubes and restraints (Score: 0-100%).Time and schedule: Orienting the patient to time and a schedule (Score: 0-100%).Home-like environment and Hearing: A comfortable environment similar to home and music (Score: 0-100%).Orientation support: assisting with a sense of person, time, and place (Score: 0-100%).Medication review : Reviewing and adjusting medications (Score: ≥20%).Early mobilization and nutrition(Score: 0-100%).
  Arms: SMART HOME Care Gruop
Combination Product: PADIS nursing intervention — pharmacological treatments for pain, agitation, delirium, immobility, and sleep disruption as well as nursing interventions
  Arms: Control Group

SUMMARY:
Background: Delirium not only has a high incidence rate among hospitalized patients but also increases mortality rates, causes distress to patients and their families, and adds to healthcare costs. Studies have shown that non-pharmacological preventive measures can effectively prevent delirium. However, critically ill patients with multiple tubes and devices cannot receive home care due to their unstable condition. Therefore, this study aims to design multiple measures resembling a home environment in the hospital ICU to reduce the incidence of delirium.

Objectives: Primary outcomes:the incidence and duration of delirium.Secondary outcomes :hospital stay, mortality rates, and patient or family satisfaction.

Methods and Procedures: A prospective randomized double-blind study design. The study is planned to be conduct from January 1,2024 to December 30,2024。 Prior to enrollment, informed consent forms will be obtained and patients from six ICUs in the hospital.

Inclusion criteria: Adult patients aged 18 or above. No maximum age limit. Patients with a Richmond Agitation-Sedation Scale score ranging from -3 to +4.Exclusion criteria: Patients with an existing diagnosis of delirium. Patients who were unable to communicate(GCS≦3）。 Patients with moderate to severe dementia.Patients with severe sedation or coma(GCS≦3）。 Sample Size: The control group's delirium incidence rate of 69.1% based on a study. The experimental group is expected to reduce delirium incidence rate to 40%。 A α value of 0.05, power 80%, each group will require 45 participants, total sample size 90 participants.A loss to follow-up rate about 15%。 To improve the effectiveness of the research design results, sample size is increased to 104 and each group is 52 participants.

Intervention Design:Each delirium assessment using the ICDSC, both groups will undergo routine assessment using RASS.

Control Group: Receive traditional comprehensive care in the ICU based on the PADIS assessment. This care will be administered by ICU nurses and will include pharmacological treatments as well as nursing interventions.

Experimental Group: ICDSC along with PRE-DELIRIC model. Intervention: In addition to the routine comprehensive care provided in the ICU, the experimental group will receive SMART HOME care interventions.

Outcome measures :ICDSC,PRE-DELIRIC,Incidence of Delirium,Duration of Delirium,LOS,Mortality Rate,Satisfaction.

DETAILED DESCRIPTION:
Prevention is better than treatment, and the intensive care unit (ICU) is a critical and highly medicalized setting where patients are prone to developing delirium. Delirium is a clinical syndrome characterized by short-term or long-term complications associated with altered consciousness and cognitive impairment. Prevention is the most crucial aspect of care, rather than waiting for it to occur and providing treatment. Delirium manifests as a rapid change in the level of consciousness and cognitive impairment. Delirium not only has a high incidence rate among hospitalized patients but also increases mortality rates, causes distress to patients and their families, and adds to healthcare costs. Studies have shown that non-pharmacological preventive measures can effectively prevent delirium. Evidence suggests that providing diverse preventive measures in the home environment of delirious patients is more effective than in a rigid hospital setting. However, critically ill patients with multiple tubes and devices cannot receive home care due to their unstable condition. Therefore, this study aims to design multiple measures resembling a home environment in the hospital ICU to reduce the incidence of delirium.

This study focuses on the ICU departments , comprising a total of six units with 72 ICU beds. The Intensive Care Delirium Screening Checklist (ICDSC) and the Richmond Agitation-Sedation Scale (RASS) are used for delirium assessment and evaluation of agitation, respectively. In 2023, a delirium assessments using ICDSC was conducted in the medical ICU of a medical center in Taiwan, with occurrence rates of 69.1%. However, there is currently no empirical research on delirium prevention measures in Taiwan, and delirium is associated with increased incidence and mortality rates, prolonged hospital stays, increased hospital costs, and long-term cognitive impairment after discharge. According to the recommendations of the Society of Critical Care Medicine (SCCM), antipsychotic drugs should not be routinely used to treat delirium in critically ill adults. Non-pharmacological treatment is currently an important option for delirium management. Therefore, this project aims to develop a predictive model for ICU delirium in Taiwan, which can intervene with diverse care preventive measures before delirium occurs .

The study consists of two groups: the SMART HOME group (experimental group) and the traditional care group (control group).

A prospective randomized double-blind study design will be adopted. After obtaining approval from the hospital's Institutional Review Board (IRB), the study is planned to be conducted from January 1,2024 to December 30,2024。 Prior to enrollment, informed consent forms will be obtained from all eligible patients or their family members (for patients who are still unconscious or unable to sign the consent form)。 The study will enroll patients from the ICU departments of six units in the hospital.

The control group will have a projected delirium incidence rate of 69.1% based on a study. The experimental group is expected to reduce the delirium incidence rate to 40%。 A α value of 0.05, and a desired power of 80%, each group will require 45 participants, resulting in a total sample size of 90 participants.A loss to follow-up rate estimated at 15%。 In order to improve the effectiveness of the research design results, the total sample size is increased to 104 people .

Prior to each delirium assessment using the ICDSC, both groups will undergo routine sedation level assessment using the RASS to evaluate their level of arousal.

The control group will use the ICDSC currently used in the hospital's ICU. The ICDSC is assesses the symptoms or fluctuations in the past 8 or 24 hours: change in consciousness, inattention, disorientation, hallucination or delusion, psychomotor agitation or retardation, inappropriate speech or mood, sleep/wake cycle disturbance, and symptom fluctuations. Each symptom present is scored as one point, with a total score of ≥4 indicating the presence of delirium. The control group will receive traditional comprehensive care in the ICU based on the PADIS (pain, agitation, delirium, immobility, sleep disruption) assessment. This care will be administered by ICU nurses and will include pharmacological treatments for pain, agitation, delirium, immobility, and sleep disruption as well as nursing interventions.

The delirium assessment in the experimental group will include the ICDSC (administered by nurses) currently used in the hospital's ICU, along with the developed information system incorporates the PRE-DELIRIC model. The PRE-DELIRIC model has been externally validated in Lithuania, Argentina and Australia. The model includes ten predictive factors that are routinely recorded in medical records, such as age, APACHE II score, admission category, coma, infection, metabolic acidosis, emergency admission, blood urea nitrogen, sedative use, and 24-hour morphine dose .The PRE-DELIRIC model categorizes patients into four risk groups: low risk (0-20%）medium risk (20-40%）high risk (40-60%）and very high risk （>60%). By utilizing these risk levels, healthcare professionals can identify patients at a higher risk of developing delirium and implement appropriate preventive measures or interventions.In addition to the routine comprehensive care provided in the ICU, the experimental group will receive SMART HOME care interventions. "SMART HOME" refers to a set of interventions aimed at preventing delirium. Sleep hygiene: Providing a quiet and dim environment for at least 6 hours (earplugs, eye masks) to facilitate sleep (Score: 0-100%).Multidisciplinary collaboration: Involving a team of various specialists such as pharmacists, respiratory therapists, rehabilitation therapists, and physical therapists (Score: ≥20%).Assessment of pain/anxiety/agitation: Evaluating and assessing the levels of pain, anxiety, and agitation (Score: 0-100%).Release of tracheal tubes and restraints: Properly relieving pressure from tracheal tubes and restraints (Score: 0-100%).Time and schedule: Orienting the patient to time and providing a schedule (Score: 0-100%).Home-like environment and Hearing: Providing a comfortable environment similar to home and incorporating gentle music (Score: 0-100%).Orientation support: assisting the patient with a sense of person, time, and place (Score: 0-100%).Medication review and adjustment: Reviewing and adjusting medications as necessary (Score: ≥20%).Early mobilization and nutrition: Initiating early rehabilitation and ensuring adequate nutrition (Score: 0-100%).

The study was conducted at a medical center in northern Taiwan, specifically targeting the intensive care unit (ICU) population. The study employed a prospective, randomized, double-blind design.

ELIGIBILITY:
Inclusion Criteria:

Moderate sedation to Combative (Richmond Agitation-Sedation Scale score : -3 to +4)

Exclusion Criteria:

Delirium. GCS≦3. Moderate to severe dementia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of delirium. | From date of randomization until the date of first documented of delirium date or delirium ended date, assessed up to 6 months.
  Incidence of Delirium: Refers to the proportion of new cases of delirium occurring in the study population after admission to the ICU (assessed using intensive care delirium screening checklist , with a score >4 point indicating delirium). It is expressed as a percentage %.
The duration of delirium | From date of randomization until the date of first documented of delirium date or delirium ended date, assessed up to 6 months.
  Duration of delirium:Refers to the time from the onset to the end of delirium in the study population after admission to the ICU. The duration can be in hours, days, or longer,Like 5 hours or 7days.

SECONDARY OUTCOMES:
Length of Stay | From date of randomization until the date of first documented of discharge or date transfer out of ICU or date of death from any cause, whichever came first, assessed up to 6 months.
  Length of Stay: Refers to the total time the patients received treatment or observation in the hospital, measured in days.
mortality rates | From date of randomization until the date of first documented of discharge or date transfer out of ICU or date of death from any cause, whichever came first, assessed up to 6 months.
  Mortality Rate: Refers to the proportion of deaths that occurred within the study population during the hospital stay, expressed as a percentage %.
patient or family satisfaction | From date of randomization until the date of first documented of discharge or date transfer out of ICU or date of death from any cause, whichever came first, assessed up to 6 months.
  Patient or Family Satisfaction: The overall satisfaction with the new multidisciplinary care measures was assessed using a Likert five-point scale, ranging from strongly disagree to strongly agree, with scores ranging from 1 to 5 point.1 point means very dissatisfied,5 points means very satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Yin Hsieh, MSN, Principal Investigator — National Taiwan University Hospital